CLINICAL TRIAL: NCT02500654
Title: Peri-implantitis - Regenerative Treatment With Enamel Matrix Derivative (EMD). Clinical Effects, Microbial Profiles and Molecular Mechanisms. A Randomised Controlled Pilot Study.
Brief Title: Regenerative Surgical Treatment of Peri-implantitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Catrine Isehed (Other)
Collaborators: Umeå University (Other)
Responsible Party: Sponsor-Investigator, Catrine Isehed, DDS, periodontist, Region Gävleborg
Organization: Region Gävleborg (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CFUG 476871
Record Dates: First submitted 2015-07-15; First posted 2015-07-16 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Failure of Dental Implant Due to Infection; Infection; Inflammation; Peri-implantitis; Bacterial Infections; Bleeding of Subgingival Space; Molecular Sequence Variation; Periodontal Diseases; Mouth Diseases
Keywords: Peri-implantitis; Regenerative therapy; Surgical therapy; Enamel matrix derivative; Peri-implant microflora; Peri-implant fluid
MeSH Terms: conditions — Infections; Inflammation; Peri-Implantitis; Bacterial Infections; Periodontal Diseases; Mouth Diseases | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgery and Emdogain® (Experimental): access peri-implant surgery with Emdogain® applied after cleaning of implant surface with saline
  Interventions: Device: Emdogain®
- Surgery alone (Placebo Comparator): access peri-implant surgery and cleaning of implant surface with saline
  Interventions: Device: Surgery alone

INTERVENTIONS:
Device: Emdogain® — Surgery and Emdogain®
  Other Names: enamel matrix derivative; enamel matrix proteins
  Arms: Surgery and Emdogain®
Device: Surgery alone — Surgery alone
  Arms: Surgery alone

SUMMARY:
The purpose of the study is to evaluate if surgical treatment of peri-implantitis with enamel matrix derivative (Emdogain®, EMD) will have an additional effect on the healing outcome, changes in the peri-implant microflora and on the inflammatory response in the periimplant pocket at 12 months.

DETAILED DESCRIPTION:
This is a randomised controlled clinical trial. Recruiting 31 patient with periimplantitis at one or more implants in need for surgical treatment.

Randomisation to test group (EMD) with surgical treatment and additional application of enamel matrix derivative (Emdogain®) or surgical treatment alone in the control group (non-EMD).

Treatment of existing periodontitis performed before recruitment. Baseline examination including samples of microbiota and peri-implant fluid followed by surgical treatment. Access surgery to remove chronic inflammatory tissue and clean the implant surface from biofilm and implant stone with hand instrument and ultrasonic device with special tips for implants, followed by polishing the implant surface with a gauze, super floss and rinsing with saline. Allocation with a performed block randomisation at the stage of surgery, after cleaning of implant surface. Application of enamel matrix derivative (Emdogain®) or not, just before closure of flap. After surgery rinsing with chlorhexidine 0.2% twice a day in 6 weeks. No systemic antibiotic used in this study.

Supportive care program, including hygiene instructions and professional cleaning supragingival at implants and teeth at 2 weeks, 3, 6, 9 and 12 months after treatment.

Examination with measurements of pocket depth and bone levels at radiographs at baseline just before surgery and 12 months and prevalence of bleeding on probing, pus or recession as well as full mouth plaque score and full mouth bleeding score at 3, 6, 9 and 12 months.

Microbial sampling performed with endodontic paper points at baseline and 2 weeks after surgery as well 3, 6 and 12 months from implant site with at baseline the deepest pocket.

Sampling of the peri-implant fluid from the peri-implant pocket at baseline, 3, 6, and 12 months from implant site with at baseline the deepest pocket.

Removal of bridges performed to give accessibility at baseline examination/surgery and at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* peri-implant angular bone loss ≥3 mm, measured at radiographs
* deep pocket ≥5 mm combined with bleeding and/or pus

Exclusion Criteria:

* individuals with uncontrolled diabetes (HbA1c > 7,0%)
* individuals where prophylaxis of antibiotic is indicated
* medication with prednisolon or other anti-inflammatory drug
* medication with gingival hyperplasia known as a side effect
* systemic antibiotic intake the last 3 months

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Changes in marginal bone level at dental implant | 12 months

SECONDARY OUTCOMES:
Changes in peri-implant microflora incidence and composition | 2weeks, 3, 6, 12 months
Changes in peri-implant pocket depth | 12 months
Number of sites with bleeding on probing | 3,6, 9, 12 months
Number of sites with bacterial plaque at the implant | 3,6, 9, 12 months
Number of sites with suppuration on probing | 3,6, 9, 12 months
Number of sites with marginal gingival recession | 3,6, 9, 12 months
Full mouth plaque score | 3,6, 9, 12 months
Full mouth bleeding score | 3,6, 9, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pernilla Lundberg, Assoc. Prof, Principal Investigator — Department of Odontology, Division of Molecular Periodontology , Umeå University, Sweden, pernilla.lundberg@umu.se
Locations (1):
- Sweden, Gävle, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Derks J, Tomasi C. Peri-implant health and disease. A systematic review of current epidemiology. J Clin Periodontol. 2015 Apr;42 Suppl 16:S158-71. doi: 10.1111/jcpe.12334. PMID 25495683
- [Background] Heitz-Mayfield LJ, Lang NP. Comparative biology of chronic and aggressive periodontitis vs. peri-implantitis. Periodontol 2000. 2010 Jun;53:167-81. doi: 10.1111/j.1600-0757.2010.00348.x. PMID 20403112
- [Background] Maruyama N, Maruyama F, Takeuchi Y, Aikawa C, Izumi Y, Nakagawa I. Intraindividual variation in core microbiota in peri-implantitis and periodontitis. Sci Rep. 2014 Oct 13;4:6602. doi: 10.1038/srep06602. PMID 25308100
- [Background] Basegmez C, Yalcin S, Yalcin F, Ersanli S, Mijiritsky E. Evaluation of periimplant crevicular fluid prostaglandin E2 and matrix metalloproteinase-8 levels from health to periimplant disease status: a prospective study. Implant Dent. 2012 Aug;21(4):306-10. doi: 10.1097/ID.0b013e3182588408. PMID 22814555
- [Background] Carcuac O, Berglundh T. Composition of human peri-implantitis and periodontitis lesions. J Dent Res. 2014 Nov;93(11):1083-8. doi: 10.1177/0022034514551754. Epub 2014 Sep 26. PMID 25261052
- [Background] Holmlund A, Hanstrom L, Lerner UH. Bone resorbing activity and cytokine levels in gingival crevicular fluid before and after treatment of periodontal disease. J Clin Periodontol. 2004 Jun;31(6):475-82. doi: 10.1111/j.1600-051X.2004.00504.x. PMID 15142219
- [Background] Bosshardt DD. Biological mediators and periodontal regeneration: a review of enamel matrix proteins at the cellular and molecular levels. J Clin Periodontol. 2008 Sep;35(8 Suppl):87-105. doi: 10.1111/j.1600-051X.2008.01264.x. PMID 18724844
- [Background] Esposito M, Grusovin MG, Worthington HV. Treatment of peri-implantitis: what interventions are effective? A Cochrane systematic review. Eur J Oral Implantol. 2012;5 Suppl:S21-41. PMID 22834392
- [Background] Casati MZ, Sallum EA, Nociti FH Jr, Caffesse RG, Sallum AW. Enamel matrix derivative and bone healing after guided bone regeneration in dehiscence-type defects around implants. A histomorphometric study in dogs. J Periodontol. 2002 Jul;73(7):789-96. doi: 10.1902/jop.2002.73.7.789. PMID 12146539